CLINICAL TRIAL: NCT01948375
Title: Effect of Blinding With a New Pragmatic Placebo Needle: a Crossover Study
Brief Title: A Crossover Study on the Blinding Effect of a New Pragmatic Placebo Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2012BAI24B01-0
Record Dates: First submitted 2013-09-08; First posted 2013-09-23 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Device Ineffective
Keywords: subject blinding; placebo needle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- real needle- placebo needle (Experimental): Participants received acupuncture with real needle in the first period, and with pragmatic placebo acupuncture needle in the second period.
  Interventions: Device: real needle- placebo needle
- placebo needle - real needle (Experimental): Participants received acupuncture with pragmatic placebo needle in the first period, and with real acupuncture needle in the second period.
  Interventions: Device: placebo needle - real needle

INTERVENTIONS:
Device: real needle- placebo needle — All acupoints were needled through the pad but just pressed against the skin without penetration by pragmatic placebo needle, while through the pad and into the skin 15 mm by real needle. For each intervention, LI4 and RN12 are needled first in a supine position for 15 minutes; BL36 and BL25 are needled secondly in a prone position for another 15 minutes. After withdrawal of the needle, participants were asked to give answers on perception of skin penetration, needle sensation and acupuncture pain. Acupuncture was given every other day, three sessions for one kind of needle, six sessions in total for each subject. There was a two-day interval between the applications of two kinds of needles.
  Arms: real needle- placebo needle
Device: placebo needle - real needle — All acupoints were needled through the pad but just pressed against the skin without penetration by pragmatic placebo needle, while through the pad and into the skin 15 mm by real needle. For each intervention, LI4 and RN12 are needled first in a supine position for 15 minutes; BL36 and BL25 are needled secondly in a prone position for another 15 minutes. After withdrawal of the needle, participants were asked to give answers on perception of skin penetration, needle sensation and acupuncture pain. Acupuncture was given every other day, three sessions for one kind of needle, six sessions in total for each subject. There was a two-day interval between the applications of two kinds of needles.
  Arms: placebo needle - real needle

SUMMARY:
Placebo needle is a useful tool to assess the efficacy of acupuncture. Investigators have applied a new kind of placebo needle in large scale acupuncture clinical trials, which named as pragmatic placebo needle. Compared with other placebo needles used in acupuncture trials, this pragmatic placebo needle shows several advantages: the outlook closer to traditional acupuncture needles, no restriction to needle depth of true needle, simple to manipulate and more economical. However, its blinding effect is not yet validated. The primary objective of this trial is to validate the blinding effect of the new pragmatic placebo needle; the secondary objective is to explore factors influencing the blinding effect of the placebo needles.

DETAILED DESCRIPTION:
blinding refers to subject blinding

ELIGIBILITY:
Inclusion Criteria:

* 18-74 years old;
* with a basic capacity of listening, speaking, reading and writing in Chinese;
* volunteer to join this research and sign the informed consent.

Exclusion Criteria:

* with acute or chronic pain;
* taking analgesics or drugs inducing abnormal sensation;
* with diseases of sensory disturbance or sensory loss;
* with alcohol or drug abuse history;
* serious cardiovascular, cerebral, hepatic, renal, hematopoietic, hemorrhagic or psychiatric diseases;
* diabetes mellitus or dermatological disease;
* women in pregnancy or lactation period;
* cardiac pacemaker carrier, metal allergy or severe needle phobia.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Study Director — Guang'an Men Hospotal Affiliated to China Academy of Chinese Medical Sciences
Locations (1):
- Guang'an Men Hospotal Affiliated to China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were recruited from Guang'anmen Hospital of China Academy of Chinese Medical Sciences via poster advertisements between August 2013 and December 2013.
Groups:
- Real Needle- Placebo Needle: Participants will accept acupuncture with real acupuncture needle in the first period, and pragmatic placebo needle in the second period of the trial.
  real needle- placebo needle: Participants will accept acupuncture with real needle in the first period and pragmatic placebo needle in the second period. Acupoints are to be needled 1 cun by real needle in the first period, and pressed against the skin with no penetration by placebo needle in the second period. For each intervention, LI4 and RN12 are needled first in a supine position for 15 minutes; BL36 and BL25 are needled secondly in a prone position for another 15 minutes. After withdrawal of the needle, participants will be asked questions on skin penetration of needles, needling pain and needle sensation. The acupuncture treatment is given every other day. There are three sessions for each kind of needle, six sessions in total for each participant. There is a two-day interval between two kinds of interventions.
- Placebo Needle - Real Needle: Participants will accept acupuncture with pragmatic placebo needle in the first period, and real acupuncture needle in the second period of the trial.
  placebo needle - real needle: Participants will accept acupuncture with pragmatic placebo needle in the first period, and real needle in the second period. Acupoints will be needled with no penetration of the skin by placebo needle, while 1 cun by real acupuncture needle. For each intervention, LI4 and RN12 are needled first in a supine position for 15 minutes; BL36 and BL25 are needled secondly in a prone position for another 15 minutes. After withdrawal of the needle, participants will be asked questions on skin penetration of needles, needling pain and needle sensation. The acupuncture treatment is given every other day. There are three sessions for each kind of needle, six sessions in total for each participant. There is a two-day interval between two kinds of interventions.
Period: Overall Study
Arm/Group | Real Needle- Placebo Needle | Placebo Needle - Real Needle
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Real Needle - Placebo Needle: Participants received acupuncture with real needle in the first period, and with pragmatic placebo acupuncture needle in the second period.
  All acupoints were needled through the pad but just pressed against the skin without penetration by pragmatic placebo needle, while through the pad and into the skin 15 mm by real needle. For each intervention, LI4 and RN12 are needled first in a supine position for 15 minutes; BL36 and BL25 are needled secondly in a prone position for another 15 minutes. After withdrawal of the needle, participants were asked to give answers on perception of skin penetration, needle sensation and acupuncture pain. Acupuncture was given every other day, three sessions for one kind of needle, six sessions in total for each subject. There was a two-day interval between the applications of two kinds of needles.
- Total: Total of all reporting groups
Arm/Group | Placebo Needle - Real Needle | Real Needle - Placebo Needle | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.47 (14.54) | 48.90 (16.74) | 49.18 (15.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 11 | 30
  Male | 11 | 19 | 30
Region of Enrollment [Number; unit: participants]
  China | 30 | 30 | 60
Educational level [Number; unit: participants]
  Secondary education and the below | 14 | 16 | 30
  Tertiary education | 16 | 14 | 30
Acupuncture experience [Number; unit: participants]
  None | 7 | 8 | 15
  1-5 sessions | 13 | 7 | 20
  6-10 sessions | 0 | 2 | 2
  >10 sessions | 10 | 13 | 23
Nervousness of acupuncture [Number; unit: participants]
  No nervous | 16 | 14 | 30
  A little nervous | 7 | 7 | 14
  Very nervous | 0 | 1 | 1
  no report | 7 | 8 | 15
Acupuncture discomfort (vas) [Median (Inter-Quartile Range); unit: score] — The discomfort of acupuncture is assessed using visual analogue scale (VAS), where 0 means no discomfort, and 10 means the severest discomfort.
  A lower value represented a better outcome, which indicated that needles used induced less pain.
  score | 0.9 [0 to 2.0] | 0 [0 to 3.5] | 0 [0 to 2.0]
Familiarity with needle sensation [Number; unit: participants]
  yes | 20 | 21 | 41
  no | 3 | 1 | 4
  no response | 7 | 8 | 15
Type of needle sensation ever experienced [Number; unit: participants]
  Distention | 18 | 20 | 38
  Soreness | 16 | 17 | 33
  Pricking | 10 | 19 | 29
  Numbness | 9 | 17 | 26
Acceptability of acupuncture [Number; unit: participants]
  Very difficult to accept | 0 | 1 | 1
  A little difficult to accept | 0 | 1 | 1
  Acceptable | 10 | 10 | 20
  Easy to accept | 5 | 5 | 10
  Very easy to accept | 8 | 5 | 13
  no response | 7 | 8 | 15
Preference of acupuncture [Number; unit: participants]
  Yes | 23 | 21 | 44
  Not sure | 0 | 1 | 1
  no response | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Volunteers'Perception of Needle Penetration Between the Pragmatic Placebo Needle and Real Needle.
Description: The primary outcome was the proportion of volunteers'perception of needle penetration between the placebo needle and the real needle in the third acupuncture session in each period.
  LI4, on the dorsum of the hand, between the first and second metacarpal bones, approximately in the center of the second metacarpal bone; RN12, on the upper abdomen,4 cun above the umbilicus,on the anterior midline; BL36, on the back of the thigh,on the midpoint of the inferior gluteal crease; BL25, on the loin, 1.5 cun lateral to the lower border of the spinous process of the fourth lumbar vertebra.
Time Frame: in the third acupuncture session in each period
Measure: Number; unit: participants
Arm/Group | Placebo Needle - Real Needle | Real Needle- Placebo Needle
Number analyzed (Participants) | 30 | 30
participants
  LI4: Preferred period 1 | 1 | 0
  LI4: No preference | 29 | 30
  LI4: Preferred period 2 | 0 | 0
  RN12: Preferred period 1 | 0 | 2
  RN12: No preference | 26 | 26
  RN12: Preferred period 2 | 4 | 2
  BL25: Preferred period 1 | 2 | 4
  BL25: No preference | 26 | 26
  BL25: Preferred period 2 | 2 | 0
  BL36: Preferred period 1 | 1 | 2
  BL36: No preference | 29 | 27
  BL36: Preferred period 2 | 0 | 1
Statistical Analysis 1: Comparison: Placebo Needle - Real Needle vs Real Needle- Placebo Needle; Test type: Superiority or Other; p > 0.05, Chi-squared

2. Secondary Outcome: Southampton Needle Sensation Questionnaire-Type of Needle Sensation
Description: This questionnaire is used to collect the types and degree of needle sensation experienced by participants. Information is collected after the third acupuncture session in each period. The difference between two kinds of needles is to be analyzed.
Time Frame: in the third acupuncture session in each period
Measure: Number; unit: participants
Arm/Group | Placebo Needle - Real Needle | Real Needle- Placebo Needle
Number analyzed (Participants) | 30 | 30
participants
  Pricking：Preferred period 1 | 8 | 6
  Pricking：No preference | 20 | 17
  Pricking：Preferred period 2 | 2 | 7
  Distending：Preferred period 1 | 1 | 7
  Distending：No preference | 20 | 21
  Distending：Preferred period 2 | 9 | 2
  Soreness：Preferred period 1 | 4 | 10
  Soreness：No preference | 18 | 16
  Soreness：Preferred period 2 | 8 | 4
  Spreading：Preferred period 1 | 3 | 6
  Spreading：No preference | 24 | 20
  Spreading：Preferred period 2 | 3 | 4

3. Secondary Outcome: Southampton Needle Sensation Questionnaire-Degree of Needle Sensation
Description: The degree of needle sensation between the placebo needle and the real needle were compared.
  The data of degree of needle sensation of the placebo needle included rows 1-4,i.e,, rows of "placebo needle:no", "placebo needle: mild", "placebo needle: moderate" and "placebo needle: severe".
  The data of degree of needle sensation of the real needle included rows 5-8, i.e., rows of "real needle: no", 'real needle: mild", "real needle: moderate", and "real needle: severe".
Time Frame: in the third acupuncture session in each period
Measure: Number; unit: participants
Arm/Group | Placebo Needle - Real Needle | Real Needle- Placebo Needle
Number analyzed (Participants) | 30 | 30
participants
  Placebo needle: No | 1 | 3
  Placebo needle: Mild | 14 | 17
  Placebo needle: Moderate | 15 | 9
  Placebo needle: Severe | 0 | 1
  Real needle: No | 0 | 1
  Real needle: Mild | 11 | 12
  Real needle: Moderate | 16 | 16
  Real needle: Severe | 3 | 1
Statistical Analysis 1: Comparison: Placebo Needle - Real Needle vs Real Needle- Placebo Needle; Test type: Superiority or Other; p = 0.007, Generalized Estimating Equation — For the comparison of direct effect of placebo needle and real needle, p=0.007; Odds Ratio (OR) = 2.35, 95% CI [1.26 to 4.40]

4. Secondary Outcome: Degree of Acupuncture Pain
Description: The pain of acupuncture is assessed using visual analogue scale (VAS), where 0 means no pain, and 10 means the imaginable severest pain. The VAS value of each period is used to compare the difference of acupuncture pain between the placebo needle and the real needle.
  A lower value represented a better outcome, which indicated that needles used induced less pain.
Time Frame: in the third acupuncture session in each period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Needle - Real Needle | Real Needle- Placebo Needle
Number analyzed (Participants) | 30 | 30
units on a scale
  placobo needle | 3.02 (1.87) | 2.73 (1.41)
  real needle | 3.70 (2.22) | 3.46 (1.98)
Statistical Analysis 1: Comparison: Placebo Needle - Real Needle vs Real Needle- Placebo Needle; Test type: Superiority or Other; p = 0.006, t-test, 2 sided — for the comparison of difference of acupuncture pain in two periods between the two groups,t=-2.88, p=0.006. t=-2.88 refers to the t value of t test

5. Secondary Outcome: Acceptability of the Acupuncture Needle
Description: After the third acupuncture of each period, participants are asked to show their acceptance toward the needles with a 5-point scale: very difficult to accept, a little difficult to accept, acceptable, easy to accept, very easy to accept.
  The needle acceptability between the placebo needle and real needle are compared.
  Data of the acceptability of the placebo needle included rows 1-5, i.e., rows of "placebo needle: very difficult to accept", "placebo needle: a little difficult to accept", "placebo needle: acceptable", "placebo needle: easy to accept" and "placebo needle: very easy to accept".
  Data of the acceptability of the real needle included rows 6-10, i.e., rows of "real needle: very difficult to accept", "real needle: a little difficult to accept", "real needle: acceptable", "real needle: easy to accept" and "real needle: very easy to accept".
Time Frame: in the third acupuncture session in each period
Measure: Number; unit: participants
Arm/Group | Placebo Needle - Real Needle | Real Needle- Placebo Needle
Number analyzed (Participants) | 30 | 30
participants
  Placebo needle: very difficult to accept | 0 | 0
  Placebo needle: a little difficult to accept | 0 | 1
  Placebo needle: acceptable | 15 | 11
  Placebo needle: easy to accept | 5 | 12
  Placebo needle: very easy to accept | 10 | 6
  Real needle: very difficult to accept | 0 | 0
  Real needle: a little difficult to accept | 2 | 2
  Real needle: acceptable | 14 | 15
  Real needle: easy to accept | 8 | 8
  Real needle: very easy to accept | 6 | 5
Statistical Analysis 1: Comparison: Placebo Needle - Real Needle vs Real Needle- Placebo Needle; Test type: Superiority or Other; p = 0.048, Generalized Estimating Equation — For the comparison of direct effect of placebo needle and real needle, p=0.048; Odds Ratio (OR) = 1.63, 95% CI [1.01 to 2.64]

ADVERSE EVENTS:
Arm/Group | Real Needle- Placebo Needle | Placebo Needle - Real Needle
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes